CLINICAL TRIAL: NCT06896136
Title: Phase 1, Randomized, Placebo-Controlled, Blinded Study in Healthy Adults Challenged With Enterotoxigenic Escherichia Coli, of the Safety, Tolerability and Anti-Diarrheal Activity of VENBETA6890, an Orally Administered, Human Monoclonal IgA
Brief Title: Study in Healthy Adults Challenged With Enterotoxigenic E. Coli, of the Safety, Tolerability and Anti-Diarrheal Activity of VENBETA6890, an Orally Administered, Human Monoclonal IgA
Acronym: MBL-ETEC-21-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mark Klempner (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Pharmaron CPC, Inc. (Unknown); University of Maryland (Other)
Responsible Party: Sponsor-Investigator, Mark Klempner, Professor of Medicine, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00084264
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Diarrhea Infectious
Keywords: ETEC; Diarrhea; Oral Prophylaxis
MeSH Terms: conditions — Dysentery; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A arm 1 Investigational Product (Experimental): Arm 1 Investigational product - Venbeta
  Interventions: Drug: VENBETA6890
- Part A Arm 2 (Placebo Comparator): Part A Arm 2 Placebo
  Interventions: Drug: Placebo
- Part B Arm 2 (Placebo Comparator): Part B Arm 2 Particpants receive placebo.
  Interventions: Drug: Placebo
- Part B Arm 1 (Experimental): Part B Arm 1 Participants receive Investigational Product
  Interventions: Drug: VENBETA6890

INTERVENTIONS:
Drug: VENBETA6890 — Part A will consist of 1 sentinel dosing group of 2 subjects randomized 1:1 to receive VENBETA6890 and will evaluate VENBETA6890 at dose levels of 15 mg/kg. On Day 1, subjects will receive 15 mg/kg in the morning and a second dose of 15 mg/kg 8 - 12 h later in the outpatient clinic. On Day 2, they will receive a third dose of 15 mg/kg at approximately 8 - 12 h after the last dose on Day 1.
  Arms: Part A arm 1 Investigational Product; Part B Arm 1
Drug: Placebo — Part A Placebo (saline) will be administered at dose levels of 15 mg/kg. On Day 1, subjects will receive 15 mg/kg in the morning and a second dose of 15 mg/kg 8 - 12 h later in the outpatient clinic. On Day 2, they will receive a third dose of 15 mg/kg at approximately 8 - 12 h after the last dose on Day 1.
  Arms: Part A Arm 2; Part B Arm 2

SUMMARY:
This is a phase 1, randomized, placebo-controlled, blinded study in up to 36 healthy adults, aged 18-45 years, challenged with Enterotoxigenic Escherichia coli, evaluating the safety, tolerability and anti-diarrheal activity of VENBETA6890, an orally administered, human monoclonal IgA.

DETAILED DESCRIPTION:
Part A will consist of 1 sentinel dosing group of 2 subjects randomized 1:1 to receive VENBETA6890 or placebo and will evaluate VENBETA6890 at dose levels of 15 mg/kg. On Day 1, subjects will receive 15 mg/kg in the morning and a second dose of 15 mg/kg 8 - 12 h later in the outpatient clinic. On Day 2, they will receive a third dose of 15 mg/kg at approximately 8 - 12 h after the last dose on Day 1. The occurrence of local and systemic reactogenicity (solicited AEs) over the subsequent 7-days post-dosing will be collected; non-solicited non-serious AEs will be collected through 28-days post-dosing and serious adverse events (SAEs) will be collected through 2 months. An independent Safety Monitoring Committee (SMC) will review the cumulative 7-day safety data for the sentinel group and must approve for the study to proceed to Part B.

Part B will consist of a single inpatient cohort of up to 34 subjects who will be randomized 1:1 to receive VENBETA6890 15 mg/kg, or placebo on Day -1 at approximately 12 h pre-challenge, Day 1 at approximately 1 h pre-challenge, and Day 1 at approximately 12 h post-challenge. All subjects will be challenged with wild-type ETEC strain H10407 and will be closely monitored on the inpatient unit for ETEC diarrheal illness. Subjects will receive the 3-day course of antibiotic therapy starting on Day 6 or earlier dependent on symptoms. Discharge from the inpatient unit is contingent upon the absence of ETEC diarrheal illness, including no diarrhea and no fever, plus two sequential negative stool cultures for ETEC separated by at least 12 hours.

An SMC will review the cumulative safety data after data collected during the Day 29 visit of the inpatient challenge cohort has been compiled.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female ages 18-45 years, inclusive at screening 2. Body weight 50 to 105 kg, inclusive at screening 3. Provide written informed consent before initiation of any study procedures. 4. Willing and able to complete all study requirements, restrictions, confinement to the Research Isolation ward, visits and procedures 5. Completion of a training session and demonstration of comprehension of the protocol procedures and knowledge of ETEC-associated illness by passing a written examination (passing grade is at least 70%).

  6. Healthy as judged by the Principal Investigator (PI) and determined by medical history, physical examination, medication history, and laboratory assessments.

  7. At Screening: Normal to Grade 1 values14 for the following laboratory determinations:
  * Complete Blood Count: WBC, absolute neutrophil count (ANC), hemoglobin, and platelet count
  * IgA
  * Comprehensive Metabolic Panel: creatinine, alanine aminotransferase (ALT), and total bilirubin
  * Urine protein and urine glucose
  * Urine illicit drug (positive cannabis allowed) and serum alcohol screening
  * Willingness to comply with COVID-19 screening PCR testing prior to dosing 8. Female subjects must be of non-childbearing potential (as defined as surgically sterile or postmenopausal for more than 1 year), or if of childbearing potential must be practicing abstinence or using an effective licensed method of birth control (e.g., history of hysterectomy or tubal ligation; use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, contraceptive patches, some intrauterine devices (IUDs), cervical sponges, diaphragms, condoms with spermicidal agents; or must have a vasectomized partner) within 28-days prior to the administration of VENBETA6890 or placebo and must agree to continue such precautions for 28 days after the last dose. A woman is eligible if she is monogamous with a vasectomized male.

Male subjects with female sexual partner(s) of reproductive potential must fall into one of the following categories to qualify for enrollment:

* Documented to be surgically sterilized (defined as having successfully undergone vasectomy at least 90 days prior to Screening)
* Must agree to use a physical barrier method of contraception (e.g., a male condom) in addition to their partner's use (if partner is a WOCBP) of a birth control method from the time of Screening until 90 days after the last dose of study drug. The following methods of contraception are acceptable for use by female partners (if WOCBP) of male subjects:

  1. Oral, implantable, transdermal, injectable, or intravaginal hormonal contraception taken for at least 90 days prior to Screening
  2. Intrauterine device (IUD [copper or hormonal])
  3. Contraceptive sponge with condom Male subjects must agree not to donate sperm from the time of Check-in through 90 days after the final dose of study drug 9. Agrees to avoid live-culture yogurt and other probiotics for at least 14 days prior to the first dose of VENBETA6890 and during the study.

     10. Agrees not to participate in another clinical trial during the study period.

Exclusion Criteria:

* 1. Positive pregnancy test at Screening or within 24 h prior to VENBETA6890 or placebo dosing 2. Breastfeeding 3. Poor venous access, as defined by inability to obtain venous blood, for screening labs, after 3 venipuncture attempts 4. Abnormal vital signs, defined as:

  * Systolic BP >150 mmHg or Diastolic BP >90 mmHg
  * Resting heart rate >100 bpm
  * Temperature ≥38.0°C 5. Abnormal electrocardiogram (ECG) parameters, defined as:
  * PR>220 msec
  * QRS>120 msec
  * QTcF>450 msec for males or >460 msec for females 6. IgA deficiency 7. Evidence of current or past infection with testing for human immunodeficiency virus (HIV), hepatitis C virus (HCV) antibody, or Hepatitis B triple screening panel (Hepatitis B surface antigen, Hepatitis B surface antibody, Hepatitis B total core antibody) with confirmatory testing as indicated.

    8. Having received prior vaccines for or have had prior infection with ETEC, Heat-Labile Toxin (LT), cholera, Campylobacter, or Shigella, within the past 3 years 9. History of diarrhea during travel to a developing country within the past 3 years 10. History of chronic gastrointestinal illness, including severe dyspepsia, lactose intolerance, or another significant gastrointestinal tract disease (e.g., irritable bowel syndrome, inflammatory bowel syndrome, gastric ulcer disease) 11. Regular use (≥ once weekly) of laxatives, anti-diarrheal agents, anti-constipation agents, or antacid therapies 12. History of major gastrointestinal surgery (uncomplicated laparoscopic appendectomy or cholecystectomy >1-year prior is permitted) 13. Abnormal bowel habits, as defined by <3 stools per week or >2 stools per day in the past 6 months 14. Use of systemic antibiotics within the past 2 weeks prior to Day 1 15. Use of topical (skin), otic, or ophthalmic antibiotics is acceptable, if those doses are not expected to result in significant systemic absorption levels 16. Use of oral, parenteral or high-dose inhaled steroids within 30 days. High-dose oral or parenteral steroids is defined as ≥20 mg total daily dose, or equivalent dose of other glucocorticoids; high-dose inhaled steroids is defined as >800 μg/day of beclomethasone dipropionate or equivalent.

    17. Use of any medication which might affect immune function* within 30 days

    *Examples include anti-cancer drugs, immunomodulating monoclonal antibody therapeutics, and rheumatologic therapies 18. Diagnosis of schizophrenia or other major psychiatric disease 19. Alcohol or drug abuse within last 5 years; current smokers or use of nicotine in any form within 6 months prior to screening and until after end of study.

    20. Presence of immunosuppression, which could be due to active neoplastic disease or a history of any hematologic malignancy (excluding resolved non-melanoma skin cancers), radiation therapy, or primary or secondary immunodeficiencies 21. History of allergy to quinolone (e.g., ciprofloxacin) or sulfa drugs (e.g., trimethoprim-sulfamethoxazole) 22. Known history of seizure disorder (remote history of a childhood seizure disorder which has completely resolved is acceptable) 23. Has consumed any nutrients or drugs with known strong cytochrome P450 3A4/5 (CYP3A4/5) inhibitors or inducers or P-glycoprotein inhibitors or inducers, starting from 14 days prior to Day 1 until the completion of study procedures at the end of study 24. Another investigational medication within 60 days or 5 half-lives, whichever is longer prior to Day 1 25. Participation in an investigational device study within 60 days prior to Day 1 26. Consumption of prescription and over-the-counter medication (including topical medications), traditional Chinese medicine, or herbal medicine, vitamin, mineral, plant, and other dietary supplements within 14 days or 5 half-lives, whichever is longer, prior to Day 1 and throughout the study 27. Consumption of liquids or foods containing grapefruit or cranberry from 7 days prior to Day 1 (Part A) or Check-in (Part B) and throughout the study 28. Consumption of any food containing poppy seeds from 48 h prior to Day 1 (Part A) or Check-in (Part B) and throughout the study 29. Donation of bone marrow or peripheral stem cells within 90 days prior to Day 1 or blood or plasma within 60 days prior to Day 1 30. Participation in strenuous exercise within 72 h prior to Day 1 (Part A) or Check-in (Part B) 31. Consumption of caffeine-containing substances within 72 h prior to Day 1 (Part A) or Check-in (Part B) 32. Occupation involving the handling of ETEC, cholera, or Shigella bacteria 33. Occupation in food handling industry or care of: very young children (<2 years old), elderly (≥70 years) or immunocompromised 34. Any other criteria which, in the investigator's opinion, would compromise the safety of the study, the ability of a subject to participate, or the results of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Experience Treatment Emergent Adverse Events | up to day 60
  The number of participants who experience treatment emergent adverse events. Severity of Treatment Emergent Adverse Events (TEAEs) are determined by changes in vital signs (VS), Physical examination (PE), and routine clinical laboratory tests.
Proportion of Participants who experience treatment emergent adverse events. | up to 60 days
  Severity of Treatment Emergent Adverse Events (TEAEs) are determined by changes in vital signs (VS), Physical examination (PE), and routine clinical laboratory tests.

SECONDARY OUTCOMES:
Number of participants experiencing diarrhea after enterotoxigenic E.coli (ETEC) challenge | 120 hours post challenge
  This outcome is measuring the number of participants who experience diarrhea after ETEC challenge. DIARRHEA is defined as at least 1 loose stool (stool consistency of Grade 3 or higher per protocol definition) of ≥ 300 g or at least 2 loose stools totaling ≥ 200 g during any 48-hour period
Proportion of participants experiencing diarrhea after ETEC challenge | 120 hours post challenge
  This outcome is measuring the proportion of participants who experience diarrhea after ETEC challenge. DIARRHEA is defined as at least 1 loose stool (stool consistency of Grade 3 or higher per protocol definition) of ≥ 300 g or at least 2 loose stools totaling ≥ 200 g during any 48-hour period

OTHER OUTCOMES:
Time to onset of diarrhea following ETEC challenge | 120 hours post challenge
  Time to onset of diarrhea following ETEC challenge
Severity of diarrhea after ETEC challenge | 120 hours post challenge
  SEVERITY: Based on the highest output over the 120 hours post-challenge, diarrhea will be graded as:
  * mild (2 or more Grade 3 - 5 stools ≥200 g total within 48 h OR a single Grade 3 - 5 stool of ≥300 g);
  * moderate (cumulative Grade 3 - 5 stools of ≥1,000 g over 96 h OR Grade 3 - 5 stools of ≥400 mL/g in 24 h OR 4 - 5 Grade 3 - 5 stools in 24 h);
  * severe (cumulative Grade 3 - 5 stools of ≥ 1,000 g in 48 h OR Grade 3 - 5 stools of ≥ 800 g in 24 h OR > 5 Grade 3 - 5 stools in 24 h).

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Investigator, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- Pharmaron CPC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No